CLINICAL TRIAL: NCT03921970
Title: The Efficacy Of Ultrasound-Guided Erector Spinae Plane Block For Postoperative Analgesia Management Following Laparoscopic Sleeve Gastrectomy Surgery: A Prospective, Randomized Study
Brief Title: Ultrasound-Guided Erector Spinae Plane Block Following Laparoscopic Sleeve Gastrectomy Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no participants
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Bahadir Ciftci, Primary researcher, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Medipol Mega Hospital
Record Dates: First submitted 2019-04-15; First posted 2019-04-19 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Obesity
Keywords: Laparoscopic sleeve gastrectomy; Postoperative pain management; Erector spina plane block
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Fourty patients aged 18-65 years old with American Society of Anesthesiologists (ASA) classification I-II and scheduled for laparoscopic sleeve gastrectomy under general anesthesia will be included in this prospective randomized study. Patients with a history of bleeding diathesis, receiving anticoagulant treatment, known local anesthetics and opioid allergy, infection of the skin at the site of the needle puncture, pregnancy or lactation, and patients who do not accept the procedure will be excluded from the study. Randomization will be achieved using a randomizing computer program. Patients will be randomly divided into two groups (Group ESP = ESP group, Group C = Control group) including 20 patients each, before entering the operating room.
Who Masked: Outcomes Assessor
Masking Description: Outcomes Assessor will be blinded to the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group ESP = ESP group (Active Comparator): ESP block (Group ESP) will be performed in the preoperative block room. US probe will be placed longitudinally 2-3 cm lateral to the T7 transvers process. From superior to inferior; trapezius (upper), rhomboideus major (middle), erector spinae (lower) muscles will be visualized on the hyperechoic transverse process. The 22G, 50 mm block needle (Braun Stimuplex Ultra 360, Germany) will be inserted in a cranio caudal direction and then for correction of the needle 5 ml normal saline solution will be enjected into the erector spina muscle fascia (figure). Following confirmation of the correct position of the needle, a dose of 20 ml %0.25 bupivacaine was administered. The same procedure will be performed at the other site (totally 40 ml %0.25 bupivacaine).
  Interventions: Other: ESP block (Group ESP)
- Group C = Control group (No Intervention): Patients will be administered paracetamol 1 gr IV every 8 hours in the postoperative period. The PCA device prepared with 10 mcg/ ml fentanyl will be attached to all patients with a protocol included 20 mcg bolus without infusion dose, 20 min lockout time and 4 hour limit.

INTERVENTIONS:
Other: ESP block (Group ESP) — Patients will be administered paracetamol 1 gr IV every 8 hours in the postoperative period. The PCA device prepared with 10 mcg/ ml fentanyl will be attached to all patients with a protocol included 20 mcg bolus without infusion dose, 20 min lockout time and 4 hour limit.
  Arms: Group ESP = ESP group

SUMMARY:
Bariatric surgery has been widely used in the treatment of obesity in recent years. It has been shown to be effective in reaching the ideal weight and reducing obesity-induced comorbidities. Laparoscopic sleeve gastrectomy (LSG) is defined as the first-step bariatric surgery for patients in the high surgical risk group. It has been shown that the laparoscopic approach has lower complication rates, shorter hospital stays, and earlier mobilization compared to open surgery. However, postoperative pain management is very important because it might cause major morbidity, especially pulmonary complications in the early postoperative period. The ultrasound (US) guided erector spina plane (ESP) block is a novel interfacial plan block defined by Forero et al. at 2016. ESP block provides thoracic analgesia at T5 level and abdominal analgesia at T7-9 level. In the literature, there is not still any randomized study evaluating ESP block efficiency for postoperative analgesia management after laparoscopic sleeve gastrectomy surgery.

DETAILED DESCRIPTION:
Prospective, Randomized Study Bariatric surgery has been widely used in the treatment of obesity in recent years. It has been shown to be effective in reaching the ideal weight and reducing obesity-induced comorbidities. Laparoscopic sleeve gastrectomy (LSG) is defined as the first-step bariatric surgery for patients in the high surgical risk group. It has been shown that the laparoscopic approach has lower complication rates, shorter hospital stays, and earlier mobilization compared to open surgery. However, postoperative pain management is very important because it might cause major morbidity, especially pulmonary complications in the early postoperative period.

General recommendations for bariatric surgery include multimodal analgesia without sedatives, local analgesic infiltration, and early mobilization. Opioid analgesics are often preferred for pain management because of their strong analgesic potentials. However, opioids have undesirable adverse effects such as sedation, dizziness, constipation, nausea, vomiting, physical dependence and addiction, hyperalgesia, immunologic and hormonal dysfunction, muscle rigidity, tolerance, and respiratory depression. The morbidly obese patients treated with opioids experience increased risk for adverse effects such as atelectasis, which causes postoperative pulmonary complications, and obstructive sleep apnea, which causes hypoxemia, postoperative ileus and longer hospital stay due to nausea and vomiting. For this reason, in 2006, the American Society of Anesthesiologists (ASA) suggested minimizing or avoiding opioids during perioperative and/or postoperative pain management to the bariatric patients. Therefore, ASA recommends the use of multimodal analgesia including local anesthesia, regional anesthesia and nonsteroidal anti-inflammatory drugs (NSAIDs).

The ultrasound (US) guided erector spina plane (ESP) block is a novel interfacial plan block defined by Forero et al. at 2016. ESP block provides thoracic analgesia at T5 level and abdominal analgesia at T7-9 level. The ESP block contains a local anesthetic injection into the deep fascia of erector spinae. This area is away from the pleural and neurological structures and thus minimizes the risk of complications due to injury. Visualization of sonoanatomy with US is easy, and the spread of local anesthesic agents can be easily seen under the erector spinae muscle. Thus, analgesia occurs in several dermatomes with cephalad-caudad way. Cadaveric studies have shown that the injection spreads to the ventral and dorsal roots of the spinal nerves and creates sensory blockade in both posterior and anterolateral thorax. In the literature, it has been reported that ESP block provides effective analgesia after ventral hernia repair surgery in a randomized controlled study. In some case series and case reports it has been reported that ESP block provides effective analgesia after abdominal and bariatric surgeries. In the literature, there is not still any randomized study evaluating ESP block efficiency for postoperative analgesia management after laparoscopic sleeve gastrectomy surgery.

The aim of this study is to evaluate the efficacy of US-guided ESP block for postoperative analgesia management following laparoscopic sleeve gastrectomy. The primary aim is to compare postoperative opioid consumption and the secondary aim is to evaluate postoperative pain scores (VAS), adverse effects related with opioids (allergic reaction, nausea, vomiting).

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification I-II
* Scheduled for laparoscopic sleeve gastrectomy under general anesthesia

Exclusion Criteria:

* Bleeding diathesis
* Receiving anticoagulant treatment
* Known local anesthetics and opioid allergy
* Infection of the skin at the site of the needle puncture
* Pregnancy or lactation
* Patients who do not accept the procedure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption by the patients at postoperative 24 hours peirod | Postoperative 24 hours
  Fentanyl using

SECONDARY OUTCOMES:
Postoperative pain scores | Postoperative 24 hours period
  Postoperative pain assessment will be performed using the VAS score (0 = no pain, 10 = the most severe pain felt). The VAS scores at rest and during cough will be recorded at postoperative 0, 2, 4, 8, 16 and 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Bahadir Ciftci, Asist.Prof, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared

REFERENCES:
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Chin KJ, Malhas L, Perlas A. The Erector Spinae Plane Block Provides Visceral Abdominal Analgesia in Bariatric Surgery: A Report of 3 Cases. Reg Anesth Pain Med. 2017 May/Jun;42(3):372-376. doi: 10.1097/AAP.0000000000000581. PMID 28272292
- [Background] Chin KJ, Adhikary S, Sarwani N, Forero M. The analgesic efficacy of pre-operative bilateral erector spinae plane (ESP) blocks in patients having ventral hernia repair. Anaesthesia. 2017 Apr;72(4):452-460. doi: 10.1111/anae.13814. Epub 2017 Feb 11. PMID 28188621